CLINICAL TRIAL: NCT04396158
Title: Effect of Radioiodine Therapy on Ovarian Reserve in Female Patients With Differentiated Thyroid Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebat Allah Ahmed Askar, Lecturer of nuclear medicine, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ovarian reserve
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Insufficiency; Radiation Exposure

STUDY DESIGN:
Intervention Model Description: self controlled case series
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention (Experimental)
  Interventions: Radiation: radioactive iodine

INTERVENTIONS:
Radiation: radioactive iodine — 80-200 mCi of radioactive iodine will be given to thyroid cancer patients

SUMMARY:
Thyroid carcinoma is the most common endocrine malignancy. Surgery is the standard therapeutic approach for patients with differentiated thyroid carcinoma (DTC), followed by radioiodine (RAI) therapy if indicated. For women with DTC, the effects of RAI therapy on gonadal and reproductive function are an important consideration. This study aimed to evaluate the effects of RAI therapy on ovarian function.

ELIGIBILITY:
Inclusion Criteria:

* Female patient in childbearing period.
* Female patient with differentiated thyroid carcinoma.
* Underwent thyroidectomy.
* Candidate for radioactive iodine therapy.

Exclusion Criteria:

* • Male patients.

  * Postmenopausal female patients.
  * Female patients with undifferentiated thyroid carcinoma.
  * Pregnant female patients.
  * Lactating female patients.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Level of anti-Müllerian (AMH) hormone | 6 months
  Level of anti-Müllerian (AMH) hormone in female patients before and after radioactive iodine therapy.